CLINICAL TRIAL: NCT06063200
Title: Methylphenidate and Response to Alcohol Cues (MARA) Pilot Study
Brief Title: Methylphenidate and Response to Alcohol Cues Pilot Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB202301428
Record Dates: First submitted 2023-09-26; First posted 2023-10-02 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Use Disorder; Attention Deficit Hyperactivity Disorder
Keywords: fMRI; EEG
MeSH Terms: conditions — Alcoholism; Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- crossover 1: methylphenidate, placebo (Other): methylphenidate (single dose, oral, 20 mg, immediate release) followed by placebo (single dose, oral)
  Interventions: Drug: Methylphenidate Pill
- crossover 2: placebo, methylphenidate (Other): placebo (single dose, oral) followed by methylphenidate (single dose, oral, 20 mg, immediate release)
  Interventions: Drug: Methylphenidate Pill

INTERVENTIONS:
Drug: Methylphenidate Pill — Single encapsulated pill
  Other Names: Ritalin

SUMMARY:
The purpose of this study is to determine whether changes in attention levels related to taking a single dose of a medication called methylphenidate, also known as Ritalin, affects responses to alcohol cues. The study will observe the effects of methylphenidate or a placebo on attentional bias and craving responses to alcohol cues through fMRI, EEG, and behavioral testing. Participants will be involved in one remote and two in-person sessions.

DETAILED DESCRIPTION:
Recent studies have revealed a robust link between attentional ability and resilience against stress-related psychopathology, in general, and against alcohol use disorder (AUD) specifically. For example, self-reported attentional ability correlates with scales of psychological resilience and with lower alcohol misuse in at-risk individuals. One mechanism by which attention may relate to resilience in AUD is through its effects on alcohol cue reactivity. Exposure to alcohol cues can induce motivation to drink alcohol for those with AUD. Leveraging the high rates of co-morbidity of AUD and attention-deficit/hyperactivity disorder, this pilot study seeks to demonstrate whether experimentally enhancing attention in individuals with both AUD and attentional deficits associated with attention-deficit/hyperactivity disorder (ADHD) reduces markers of addiction severity (i.e., craving and attentional bias responses to alcohol cues) and will explore the neural and behavioral mechanisms. Methylphenidate not only improves sustained attention, but in users of cocaine and methamphetamine, it was previously shown to reduce craving, attentional bias, and neural responses to viewing drug-related cues. Here we will use this commonly-prescribed medication as a pharmacological probe of attentional processes related to alcohol use disorder. We hypothesize that acute methylphenidate-associated attentional enhancement will engage compensatory brain mechanisms that will lead to attenuated craving, reduced attentional bias, and modulated neural responses to alcohol cues in young adults with AUD and ADHD. Thirty young adults with AUD and ADHD will be recruited for a double-blind, placebo-controlled, within-subjects experiment to test the effects of an acute 20 mg MPH administration to increase attention on cue-induced alcohol craving [during simultaneous functional magnetic resonance imaging (fMRI) and EEG] and attentional bias. Subjects will also perform computerized tasks of general attention with non-alcohol-related stimuli. The goal of this project is to support the design and funding proposal of a larger study.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-25 years
* Meets DSM-5 criteria for AUD
* Meets DSM-5 criteria for ADHD
* Fluent in English
* Normal or corrected to normal vision

Exclusion Criteria:

* Meets DSM-5 criteria for bipolar disorder, psychotic disorders, neurological disorders, or substance use disorders other than AUD.
* Participant routinely uses psychoactive drugs or medications except for non-dependent marijuana or nicotine use (due to common use of these substances in individuals with AUD).
* Participant has contraindications for taking methylphenidate.
* Participant has contraindications for being in an MRI machine
* Self-reported history of high blood pressure over 140/90 or consistent readings of 140/90 or above upon arrival for a session.
* History of seizure disorder
* Liver disease
* Participant is currently pregnant or trying to become pregnant

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Neural responses to cues | 15 minutes
  Cue-elicited EEG and fMRI responses. We will contrast brain activation following alcohol images with brain activation following neutral images.
Self-reported craving | 15 minutes
  Craving following presentation of alcohol and neutral images will be reported using 0-10 visual analog scales. We will contrast craving following the alcohol images with craving following the neutral images.
Accuracy on the attentional blink task | 5 minutes
  We will contrast accuracy during alcohol distractor trials with neutral distractor trials for "lags" of 8 versus 2 images following the distractor.

SECONDARY OUTCOMES:
Self-reported anxiety | 15 minutes
  Anxiety following presentation of alcohol and neutral images will be reported using 0-10 visual analog scales. We will contrast anxiety following the alcohol images with anxiety following the neutral images.
Continuous performance task omission errors | 5 minutes
  Total number of omission errors, indexing sustained attention
Attention network task reaction times | 15 minutes
  response time (RT) difference for no cue vs. central cue ("altering"), RT difference for central cue vs. spatial cue ("orienting"), RT difference for incongruent vs. congruent flankers ("executive control")
Heart rate | 15 minutes
  Heart rate will be recorded during cue-induced craving. We will contrast heart rate during the alcohol images and heart rate during the neutral images.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States